CLINICAL TRIAL: NCT05987215
Title: Interest of Using Deep Learning Algorithm for Otosclerosis Detection on Temporal Bone High Resolution CT
Acronym: OtoIA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 22-5019 / 69HCL22_1193
Record Dates: First submitted 2023-05-17; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-05

CONDITIONS: Otosclerosis
Keywords: otosclerosis; IA; deep learning; temporal bone CT
MeSH Terms: conditions — Otosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CASE: Patients with surgically confirmed otosclerosis who initially consulted for conductive hearing loss with normal otoscopy, and with a high resolution computed tomography of temporal bone available
  Interventions: Combination Product: Radiologic diagnosis; Diagnostic Test: Artificial intelligence diagnosis
- CONTROL: Random patients with a high resolution computed tomography scan of temporal bone performed without suspicion of otosclerosis and considered normal
  Interventions: Combination Product: Radiologic diagnosis; Diagnostic Test: Artificial intelligence diagnosis

INTERVENTIONS:
Combination Product: Radiologic diagnosis — Each CT scan is interpreted by a radiologist and is assigned as positive or negative for the diagnosis of otosclerosis
Diagnostic Test: Artificial intelligence diagnosis — Each CT scan is screened by the deep learning algorithm and is assigned as positive or negative for the diagnosis of otosclerosis

SUMMARY:
Otosclerosis is a relatively frequent pathology, of multifactorial origin with genetic and hormonal part, predominantly in women. This disease causes a disorder of the bone metabolism of the middle and inner ear, responsible for a progressive deafness, which can become severe.

Several elements are necessary to make the diagnosis of otosclerosis: the clinical examination and questioning, the audiometric assessment, and finally the temporal bone CT.

The CT scan allows to detect foci of otosclerosis within the bone of the middle or inner ear. This diagnosis is sometimes difficult and requires interpretation by a trained radiologist.

The investigators would like to evaluate the ability of a deep learning algorithm to detect these foci of otosclerosis, and to compare its diagnostic performance with a trained radiologist.

DETAILED DESCRIPTION:
Otosclerosis is a relatively frequent pathology, of multifactorial origin with genetic and hormonal part, predominantly in women. This disease causes a disorder of the bone metabolism of the middle and inner ear, responsible for a progressive deafness, which can become severe.

Several elements are necessary to make the diagnosis of otosclerosis: the clinical examination and questioning, the audiometric assessment, and finally the temporal bone CT.

The CT scan allows to detect foci of otosclerosis within the bone of the middle or inner ear. This diagnosis is sometimes difficult and requires interpretation by a trained radiologist.

The investigators would like to evaluate the ability of a deep learning algorithm to detect these foci of otosclerosis, and to compare its diagnostic performance with a trained radiologist.

ELIGIBILITY:
* Inclusion Criteria * :

  * age over 18
  * high resolution temporal bone CT scan available for analysis
  * for the "case" group : surgical confirmation of positive diagnosis for otosclerosis
  * for the "control" group : a first radiological analysis in favor of a normal temporal bone CT scanner and an initial radiologic report considered normal as well
* Exclusion Criteria * :

  * age under 18
  * no high resolution temporal bone CT scan available for analysis
  * unwillingness to participate in the study

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include cases from a group of patients who have undergone surgery for otosclerosis at the Lyon Sud hospital in France, and controls who have had a high resolution temporal bone CT scan at the Lyon Sud hospital with no clinical suspicion for otosclerosis and considered normal.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of the artificial intelligence algorithm compared to the diagnostic performance of the radiologist : sensitivity, specificity, positive and negative predictive value, area under the ROC curve | through study completion, an average of 5 months
  These diagnostic performances will be established from the positive or negative diagnoses of the algorithm and the radiologist, compared to the "case" or "control" status of each patient included in the study

CONTACTS AND LOCATIONS:
Overall Officials: Maxime FIEUX, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Centre Hospitalier Lyon sud, Service d'ORL, d'otoneurchirurgie et de chirurgie cervico-facaile, Pierre-Bénite, France